CLINICAL TRIAL: NCT04534699
Title: A Phase 1, Open Label, Nonrandomized, Single-dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of KBP-5074 in Subjects With Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics of KBP-5074 in Patients With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBP5074-1-006
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Moderate Hepatic Impairment; Healthy
Keywords: Hepatic Impairment; Moderate Hepatic Impairment; Healthy; KBP-5074
MeSH Terms: interventions — KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hepatic Impaired (Experimental): KBP-5074 0.5mg tablet orally, Single dose
  Interventions: Drug: KBP-5074
- Matched-control Healthy (Experimental): KBP-5074 0.5mg tablet orally, Single dose
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: KBP-5074 — KBP-5074 tablet

SUMMARY:
This multiple-center, nonrandomized, open label, parallel group, single dose study will be conducted in male and female subjects with normal hepatic function or moderate (Child-Pugh Class B) hepatic impairment to evaluate the effect of hepatic impairment on the pharmacokinetics (PK) of KBP-5074.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females, of any race, between 18 and 80 years of age, inclusive, at screening.
2. Body mass index between 18.0 and 40.0 kg/m2, inclusive, at screening.
3. Subjects with normal hepatic function must be in good health.
4. Subjects must meet the criteria for moderate hepatic impairment based on Child Pugh B.

Key Exclusion Criteria:

1. Significant history or clinical manifestation of any medical history, as determined by the investigator not appropriate to participate in this study.
2. Positive serology test results for hepatitis B surface antigen and/or human immunodeficiency virus 1/2.
3. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to dosing, whichever is longer.
4. Use of mineralocorticoids or MRAs (eg, spironolactone or eplenerone) within 90 days prior to study drug administration, unless deemed acceptable by the medical monitor and sponsor.
5. Subject has used prescription drugs within 30 days of study drug administration, with the exception of established therapy for hepatic disease and the treatment of associated disorders that have been stable for at least 30 days before study drug administration, as approved by the investigator and in consultation with the medical monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Maximum observed concentration (Cmax) | 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 264 hours postdose.
  Maximum observed concentration (Cmax) - Plasma
Pharmacokinetic Paramete: Area under the concentration-time curve from time 0 to infinity (AUC0-∞) | 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 264 hours postdose.
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) - Plasma
Pharmacokinetic Parameter: Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) | 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 264 hours postdose.
  Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) - Plasma
Pharmacokinetic Parameter: Time of the maximum observed concentration (tmax) | 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, and 264 hours postdose.
  Time of the maximum observed concentration (tmax) - Plasma
Safety of KBP-5074 by assessing the number of adverse events, laboratory abnormalities, ECGs, vital signs and physical examinations | Up to 12 days
  Incidence of severity of AEs, laboratory abnormalities (based on hematology, clinical chemistry, and urinalysis test results), ECGs, vital signs, and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: James McCabe, Study Director — KBP Biosciences
Locations (3):
- United States (3):
  - Orlando Clinical Research Center (OCRC), Orlando, Florida
  - Texas Liver Institute (TLI), San Antonio, Texas
  - Clinical Trials of Texas (CTT), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCabe J, Zhang J, Yang F, Benn V. Pharmacokinetics of the Novel Nonsteroidal Mineralocorticoid Receptor Antagonist Ocedurenone (KBP-5074) in Individuals with Moderate Hepatic Impairment. Eur J Drug Metab Pharmacokinet. 2024 Mar;49(2):229-237. doi: 10.1007/s13318-024-00879-3. Epub 2024 Feb 8. PMID 38329646